CLINICAL TRIAL: NCT03028285
Title: Open Randomized Study of the Safety, Tolerability, and Pharmacokinetic Parameters of UNIFUZOL® (Solution for Infusions, 1.4%, Manufactured by "NTFF"POLYSAN " Ltd.,Russia) in Healthy Volunteers at Different Rates of Administration (Phase I)
Brief Title: Study of Safety and Tolerability of UNIFUZOL (Solution for Infusions) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNI-I-2015
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Vascular Disease
Keywords: succinate; arginine; vasodilation; peripheral vascular disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unifusol 250 ml IV, 3 ml/mil (Experimental): Twelve healthy volunteers will receive the experimental drug (arginine sodium succinate 1.4% solution; Unifusol) intravenously at a dose 250 ml and infusion rate 3 ml/min.
  Interventions: Drug: arginine sodium succinate
- Unifusol 250 ml IV, 4.5 ml/min (Experimental): Twenty-four healthy volunteers will receive arginine sodium succinate 1.4% solution (Unifusol) intravenously at a dose 250 ml and infusion rate 4.5 ml/min
  Interventions: Drug: arginine sodium succinate
- Unifusol 500 ml IV, 4.5 ml/min (Experimental): Twelve healthy volunteers will receive arginine sodium succinate 1.4% solution (Unifusol) intravenously at a dose 500 ml and infusion rate 4.5 ml/min
  Interventions: Drug: arginine sodium succinate

INTERVENTIONS:
Drug: arginine sodium succinate — Healthy volunteers will receive the experimental drug (arginine sodium succinate 1.4% solution; Unifusol) intravenously at 3 different combinations of dose and infusion rate under the close monitoring of vital signs and other safety parameters.
  Other Names: Unifusol

SUMMARY:
Unifusol (R) is a solution of arginine sodium succinate for intravenous infusions. Its effects include vasodilation, protection of inner layer of blood vessels and improvement of blood viscosity. The present phase I study is aimed to evaluate the safety and tolerability of Unifusol infusions in healthy volunteers.

DETAILED DESCRIPTION:
Unifuzol, solution for infusions,("NTFF POLYSAN" Ltd., Russia) contains succinic acid and arginine as active ingredients; it has demonstrated cardioprotective, anti-ischemic, endothelial protective and fibrinolytic activity in pre-clinical studies and is considered for clinical trials in peripheral vascular disease.

The primary aim of the present Phase I study is to assess safety and tolerability of Unifusol (1.4% solution for infusions) at different infusion rates in healthy volunteers.

Study objectives:

1. Assess the safety parameters (vital signs, the incidence of AEs, SAEs, laboratory abnormalities) during infusion of Unifusol (1.4% solution for infusions) in healthy volunteers at different infusion rates.

   * administration of a single infusion of 250 ml at a rate of 3 ml / min.
   * administration of a single infusion of 250 ml at a rate of 4.5 ml / min
   * administration of a single infusion of 500 ml at a rate of 4.5 ml / min
2. Study the pharmacokinetics parameters of the active components of the Unifusol (succinic acid and arginine) in healthy volunteers after single infusion at a dose of 250 ml at a rate of 4.5 ml / min.

Study methods:

1. Determination of pharmacokinetic parameters of succinic acid administered at a single Unifusol infusion dose 250 ml at a rate of 4.5 ml / min (AUC, Cmax, Tmax, T1 / 2);
2. Determination of pharmacokinetic parameters of arginine after a single Unifusol infusion at a dose 250 ml at a rate of 4.5 ml / min (AUC, Cmax, Tmax, T1 / 2);
3. Determination of individual variations of the pharmacokinetic parameters of succinic acid and arginine in healthy volunteers;
4. Identification of significant gender differences in the pharmacokinetics of the active ingredients of Unifusol (succinic acid and arginine) in healthy volunteers;
5. Determination of the number of compartments in the pharmacokinetic model which will be most appropriate to the measured concentrations after a single infusion (single-chamber, two-chamber or three-chamber pharmacokinetic model).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy condition, as verified by standard clinical, laboratory and instrumental methods of examination.
2. The body mass index (BMI) of 18.5 to 30 and a body weight above 50 kg.
3. Signed informed consent.
4. For men - consent to use the double-barrier contraceptive method during the course of the study, and for 90 days after the study completion.
5. For women - negative pregnancy test, absence of lactation, and consent to use the double-barrier method of contraception during the study and for 90 days after study completion. In the case of hormonal contraceptive use, the intake must be canceled no later than 2 months before the start of the study.

Exclusion Criteria:

1. Intolerance or hypersensitivity to the components of the study drug.
2. Chronic diseases of the cardiovascular, bronchopulmonary (including bronchospastic disease), neuroendocrine system, chronic diseases of the gastrointestinal tract, liver, kidneys, blood, immune system, mental illness or substance abuse, or a history of alcoholism.
3. Acute infectious diseases within 4 weeks before the start of the study.
4. Any abnormalities of the laboratory findings before inclusion.
5. The presence of mental disorders, or the history of mental illness.\
6. Intake of medications and/or nutritional supplements for 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug, or using drugs that have a significant effect on hemodynamics, liver function, etc. (for instance, barbiturates, omeprazole, cimetidine) for 2 months prior to the first dose of study medication. Receiving herbal medicines and herbal supplements during the 28 days before the first dose of study medication.
7. Hormonal methods of contraception with systemic effects (including oral and transdermal contraceptives, injectable progesterone, subcutaneous implants with a progestin intrauterine device with progesterone release) and hormone replacement therapy within 60 days prior to the first dose of study medication.
8. The injection of any drug, depot (slow release) or the use of drug implant within 3 months prior to the administration of the study drug.
9. Abnormalities of vital signs: systolic blood pressure below 100 mm Hg or higher than 130 mm Hg; diastolic blood pressure below 60 mmHg or above 90 mm Hg; heart rate below 60 beats / min or above 90 beats / min.
10. Data of 12-lead ECG demonstrating the QTc interval> 450 msec or the QRS> 120 ms on screening visit.
11. Blood donation (450 ml of blood or more) in less than 3 months prior to inclusion.
12. Participation in clinical trials of drugs in 3 months before inclusion.
13. The regular consumption of more than 5 units of alcohol per week (each unit is equal to 30 ml of ethanol or 325 ml of beer) or the history of alcoholism, drug addiction, drug abuse.
14. A positive test for alcohol in the exhaled air.
15. Smoking more than 10 cigarettes per day.
16. A positive urine test for drugs, such as amphetamine, marijuana, morphine, cocaine and methamphetamine, and tricyclic antidepressants, as revealed in urine by immunoassay analysis.
17. The positive results of the analyzes for hepatitis B or C, HIV, and/or syphilis.
18. Unwilling or unable to give up alcohol intake, smoking and excessive exercise 48 hours prior to study drug administration and up to 96 hours after administration of the drug, as well as food and beverages containing methylxanthines and grapefruit / grapefruit juice from the day prior to the screening visit and at follow-up.
19. Compliance to a special diet (eg. vegetarian) or lifestyle (including night work and extreme exercise, such as sports or weight lifting) that may interfere with the study procedures.
20. Planning inpatient treatment of the volunteer within one month after the first injection of the study drug.
21. Lack of intention to comply with the study regimen.
22. Obvious or probable inability of volunteer, according to the judgement of the researcher, to understand and evaluate information about the study and consciously sign the informed consent form, in particular with respect to the expected risks and possible discomfort.
23. Expected problem with the placement of venous catheters or performing vein puncture.
24. Pregnancy or breast-feeding; unwillingness or inability of a woman of childbearing age to use acceptable methods of barrier contraception, according to the protocol, starting at least 14 days prior to the first dose of study medication and for 90 days after study completion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events, derangements of vital signs, and laboratory abnormalities | 18-26 days
  Absence of vital disorders, SAEs, laboratory abnormalities, and the incidence of AEs

SECONDARY OUTCOMES:
Area under the plasma concentration of arginine versus time curve | 6 hours
  AUC
Area under the plasma concentration of succinic acid versus time curve | 6 hours
  AUC
Peak Plasma Concentration of arginine | 6 hours
  Cmax
Peak Plasma Concentration of succinic acid | 6 hours
  Cmax
Time to peak Plasma Concentration of arginine | 6 hours
  Tmax
Time to peak Plasma Concentration of succinic acid | 6 hours
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Vasily B Vasilyuk, MD, PhD, Principal Investigator — Research Center for Eco-safety
Locations (2):
- Russia (2):
  - Clinical diagnostic laboratory of City Clinical Hospital named after I.V.Davydovsky, Moscow
  - Research Center for Eco-safety, Ltd., Saint Petersburg

IPD SHARING:
Plan to Share IPD: No